CLINICAL TRIAL: NCT03505489
Title: The Effect of Deep Inhalation on Mannitol Responsiveness
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Don Cockcroft, Professor, College of Medicine, University of Saskatchewan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MAN-2018
Record Dates: First submitted 2018-03-29; First posted 2018-04-23 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Asthma
Keywords: Mannitol; Methacholine; Deep inhalation; Tidal breathing
MeSH Terms: conditions — Asthma | interventions — Methacholine Chloride; Mannitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mannitol challenge (Experimental): Mannitol challenge performed per standard mannitol challenge procedure with deep inhalation technique
  Interventions: Procedure: Deep inhalation technique; Drug: Mannitol
- Mannitol challenge w/ TBI (Experimental): Mannitol challenge performed per standard mannitol challenge procedure except with tidal breathing technique
  Interventions: Procedure: Tidal breathing technique; Drug: Mannitol
- Methacholine challenge w/ DI (Experimental): Methacholine challenge performed per standard 2-minute tidal breathing challenge procedure except with deep inhalation technique
  Interventions: Procedure: Deep inhalation technique; Drug: Methacholine
- Methacholine challenge (Experimental): Methacholine challenge performed per standard 2-minute tidal breathing challenge procedure (tidal breathing technique)
  Interventions: Procedure: Tidal breathing technique; Drug: Methacholine

INTERVENTIONS:
Procedure: Deep inhalation technique — Use of deep inhalations for administration of inhalant
  Arms: Mannitol challenge; Methacholine challenge w/ DI
Procedure: Tidal breathing technique — Use of tidal breathing for administration of inhalant
  Arms: Mannitol challenge w/ TBI; Methacholine challenge
Drug: Methacholine — Methacholine direct bronchoconstrictor used for bronchoprovocation challenge
  Other Names: Provocholine
  Arms: Methacholine challenge; Methacholine challenge w/ DI
Drug: Mannitol — Mannitol indirect bronchoconstrictor used for bronchoprovocation challenge
  Other Names: Aridol
  Arms: Mannitol challenge; Mannitol challenge w/ TBI

SUMMARY:
The study will assess how the inhalation technique used (deep inhalations versus tidal breathing) influences the results of a mannitol challenge test and a methacholine challenge test, if at all.

DETAILED DESCRIPTION:
This study will look at airway responsiveness to inhaled methacholine and mannitol administered with and without deep inhalation. This study will also investigate the role of airway inflammation on these responses, using sputum differential cell counts and fractional exhaled nitric oxide.

This is a single center, open label, randomized study. Individuals with stable asthma will be eligible for enrollment. The study will consist of two parts, screening and testing.

Part 1: Screening

Participants will undergo consent procedures and assessments of fractional exhaled nitric oxide levels, airway responsiveness to methacholine and sputum induction. If participants show airway responsiveness to methacholine (i.e. methacholine PC20 16mg/mL), they will be scheduled to undergo the testing part of the study.

Part 2: Testing

Participants will be randomized to undergo two methacholine or two mannitol challenges. Further randomization will occur with respect to whether the standard challenge method or the modified challenge method is performed first.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* men and women between 18 and 75 years of age
* FEV1 at first measurement of greater than or equal to 65% predicted
* methacholine provocative concentration causing a 20% in FEV1 at screening that is less than or equal to 16mg/ml
* generally good health
* stable asthma

Exclusion Criteria:

* respiratory infection within 4 weeks of screening visit
* worsening of asthma within 4 weeks of screening visit
* lung disease other than asthma
* significant medical comorbidity
* current smoker or ex-smoker with significant smoking history
* currently pregnant or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Effect of deep inhalation (versus tidal breathing) on mannitol provocative dose causing a 15% fall in forced expiratory volume in one second (FEV1) | 24 hours between mannitol challenges
  Shift in mannitol provocative dose causing a 15% fall in forced expiratory volume

SECONDARY OUTCOMES:
Effect of airway inflammation on methacholine and mannitol challenge results-fractional exhaled nitric oxide | up to 2 weeks, from baseline to end of study
  Collection of fractional exhaled nitric oxide at screening - analysis of resulting measurement indicative of degree of baseline airway inflammation
Effect of airway inflammation on methacholine and mannitol challenge results-sputum | up to 2 weeks, from baseline to end of study
  Collection of sputum at screening - analysis for differential cell counts indicative of degree of baseline airway inflammation
Effect of deep inhalation (versus tidal breathing) on methacholine provocative | 24 hours between methacholine challenges
  Shift in methacholine provocative dose causing a 20% fall in forced expiratory volume

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Don Cockcroft, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- Asthma Research Lab - University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blais CM, Davis BE, Cockcroft DW. The effect of deep inhalation on mannitol responsiveness. Clin Exp Allergy. 2020 Mar;50(3):308-314. doi: 10.1111/cea.13543. Epub 2019 Dec 14. PMID 31785175
- [Derived] Blais CM, Davis BE, Graham BL, Cockcroft DW. Respiratory Duty Cycles in Individuals With and Without Airway Hyperresponsiveness. Chest. 2020 Feb;157(2):356-362. doi: 10.1016/j.chest.2019.09.005. Epub 2019 Sep 19. PMID 31542451